CLINICAL TRIAL: NCT07091435
Title: ChatGPT -Based Intervention for Social Frailty in Older Women With CHF : Gender Differences, Predictive Modeling, and Longitudinal Evaluation
Brief Title: ChatGPT -Based Intervention for Social Frailty in Older Women With CHF : Gender Differences
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, WANG, JENG, Professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202500678B0
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: 65 Years Older; CHF - Congestive Heart Failure; Social Communication
Keywords: older women; social frailty; CHF
MeSH Terms: conditions — Heart Failure; Communication | interventions — Community Psychiatry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention)
- ChatGPT intervention (Experimental)
  Interventions: Behavioral: ChatGPT
- Community social participation group (Experimental)
  Interventions: Behavioral: community social

INTERVENTIONS:
Behavioral: ChatGPT — Phase 2 Involves a quasi-experimental design with 174 participants identified as having low social frailty scores, randomly assigned to one of three groups: a ChatGPT intervention group engaging in daily 15-30-minute app-based conversations with emotional monitoring; a community social participation group attending regular social activities; and a control group maintaining routine activities. Outcomes related to emotional state, physical activity, social frailty, and prognosis will be assessed pre- and post-intervention.
  Arms: ChatGPT intervention
Behavioral: community social — Phase 2 involves a quasi-experimental design with 174 participants identified as having low social frailty scores, randomly assigned to one of three groups: a ChatGPT intervention group engaging in daily 15-30-minute app-based conversations with emotional monitoring; a community social participation group attending regular social activities; and a control group maintaining routine activities. Outcomes related to emotional state, physical activity, social frailty, and prognosis will be assessed pre- and post-intervention.
  Arms: Community social participation group

SUMMARY:
The study is planned to be completed over three years and will focus on 500 hospitalized older adults with a diagnosis of CHF. The Biopsychosocial model will be used to conduct this study. Phase 1: This phase aims to determine the incidence rates of sarcopenia, frailty/social frailty among hospitalized older adults, and to compare these outcomes in gender differences. Sarcopenia will be identified according to the AWGS guidelines, while clinical characteristics, including ejection fraction, stage of CHF, and comorbidities, will be collected via chart review using the 2024 Guidelines of the Taiwan Society of Cardiology(Y. H. Li et al., 2024). Frailty and social frailty will be measured using the CFS, Tilburg Frailty Indicator (TFI), and Makizako's Social Frailty Questionnaire, respectively, and physical activity levels will be assessed with the International Physical Activity Questionnaire - Short Form (IPAQ-S). To develop a predictive model examining risk factors for social frailty and health outcomes, with a focus on gender differences, we will employ Structural Equation Modeling (SEM). SEM allows for the analysis of complex relationships among variables, facilitating a comprehensive understanding of how these factors interact differently across genders. Phase 2: A quasi-experimental design will be implemented, involving 174 hospitalized older adults with low social frailty scores. Participants will be randomly assigned to one of three groups. Group 1 will use the ChatGPT app for 15-30 minutes daily, with the app actively monitoring their emotional status and automatically notifying the research team and family members if signs of negative mood are detected. Group 2 will be encouraged to increase their social participation through community-based activities. The Control Group will continue their routine lifestyle without additional interventions. Before the intervention, one-on-one training will be provided to Group 1 participants on how to use ChatGPT. Key outcome measures, including mood status (loneliness, anxiety, and depression), physical activity (assessed via IPAQ-S), overall frailty (CFS & TFI), social frailty scores, and other health indicators, will be assessed at baseline and immediately post-intervention. Phase 3: The aim of this phase is to monitor and compare the longitudinal health outcomes of interventions among the three groups. Key health outcomes will be assessed and compared every three months over a one-year period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 65 years or older.
* Diagnosis of CHF with a left ventricular ejection fraction (EF) of less than 40%
* Ability to communicate effectively in Mandarin or Taiwanese.

Exclusion Criteria:

* Patients diagnosed with unstable heart failure
* Severe Comorbidities, conditions such as end-stage renal disease, advanced hepatic dysfunction, or terminal malignancies.
* Severe cognitive deficits that impede the ability to provide informed consent or participate in study interventions.
* Uncorrected visual or hearing impairments that would hinder effective communication or interaction with the ChatGPT application.
* Active psychiatric conditions, including major depression or psychosis, that could interfere with study participation or adherence.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Tilburg Frailty Indicator (TFI) | Baseline, 3-month follow-up,6-month follow-up,12-month follow-up
  Assesses multidimensional frailty across physical, psychological, and social domains using a 15-item questionnaire. It consists of two parts: the first part gathers data on determinants of frailty (e.g., age, gender, marital status), while the second part includes 15 items divided into physical (8 items), psychological (4 items), and social (3 items) domains. This instrument offers a holistic view of an individual's frailty status. The TFI has shown good internal consistency (Cronbach's α = 0.79) and predictive validity for adverse outcomes, including functional decline and mortality Score range : 0-15 Scores 0-4 Scores: non-frail ; 5 Scores or more: frail
Makizako Social Frailty Index | Baseline, 3-month follow-up,6-month follow-up,12-month follow-up
  Assesses social frailty through a set of 5 questions related to social participation, activities, and support networks. The questionnaire has demonstrated good test-retest reliability and criterion validity in predicting adverse health outcomes such as reduced physical activity and functional decline. These instruments collectively provide a comprehensive framework for assessing physical, psychological, and social frailty, especially in studies involving older adults.
  Score range : 0-5 Scores 0 Scores: non-Social Frailty ;
  1. Scores : Pre-Social Frailty ;
  2. Scores or more: Social Frailty
International Physical Activity Questionnaire - Short Form (IPAQ-S) | Baseline, 3-month follow-up,6-month follow-up,12-month follow-up
  A self-reported measure assessing physical activity over the last seven days. It categorizes activity levels based on frequency and intensity, covering domains such as walking, moderate activity, and vigorous activity.
  Calculate MET-minutes/week Category 1: Low No activity is reported & Activity does not meet the criteria for Moderate or High categories.
  Category 2: Moderate
  Meets any of the following:
  3 or more days of vigorous activity of at least 20 min/day ; 5 or more days of moderate activity and/or walking of at least 30 min/day ; 5 or more days of any combination of walking, moderate, or vigorous activities, achieving at least 600 MET-min/week Category 3: Vigorous
  Meets either of the following:
  At least 3 days, accumulating at least 1500 MET-min/week, OR 7 or more days of any combination of activities totaling ≥3000 MET-min/week
Minnesota Living with Heart Failure Questionnaire（MLHFQ） | Baseline, 3-month follow-up,6-month follow-up,12-month follow-up
  One of the most widely used health-related quality of life questionnaires for patients with CHF.
  Score range : 0-105 Scores 0-24 Scores: Low impact of heart failure on life ; 25-45 Scores: Moderate impact of heart failure on life ; 46 Scores or more: Serious impact of heart failure on life
UCLA Loneliness Scale | Baseline, 3-month follow-up,6-month follow-up,12-month follow-up
  Measures subjective feelings of loneliness and social isolation. Score range : 6-18 Scores Higher total scores indicate greater feelings of loneliness.
Geriatric Depression Scale (GDS-15) | Baseline, 3-month follow-up,6-month follow-up,12-month follow-up
  A shorter 15-item version and designed to screen for depression in older adults.
  Scoring :
  Each depressive answer scores 1 point. Some items count "Yes" as a point. Some items count "No" as a point. The maximum total score is 15. Items Scored as 1 Point for a "Yes" Answer:1, 5, 7, 11, 13 Items Scored as 1 Point for a "No" Answer:2, 3, 4, 6, 8, 9, 10, 12, 14, 15 Interpretation of Scores 0-6: Normal (no depression) ; 7-10: Moderate depression ; 11-15: Severe depression
Clinical Frailty Scale (CFS) | Baseline, 3-month follow-up,6-month follow-up,12-month follow-up
  A 9-point scale that evaluates an individual's level of frailty based on their physical functioning and overall health status.
  Scoring Range :
  The scale ranges from 1 to 9, with higher scores indicating greater frailty.

IPD SHARING:
Plan to Share IPD: No